CLINICAL TRIAL: NCT04762095
Title: The Effect of Mindfulness Stress Reduction Program on Menopausal Complaints and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NURDİLAN SENER (Other)
Responsible Party: Sponsor-Investigator, NURDİLAN SENER, phd research assistant, Firat University
Organization: Firat University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Firat
Record Dates: First submitted 2021-02-13; First posted 2021-02-21 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Postmenopausal Women

STUDY DESIGN:
Intervention Model Description: Research is quasi-experimental
Who Masked: Participant
Masking Description: Postmenopausal Women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of mindfulness stress reduction program Quality of Life (Experimental): mindfulness stress reduction program reduces menopausal complaints.
  Interventions: Other: mindfulness stress reduction program
- The Effect of mindfulness stress reduction program Menopausal Symptoms (Experimental): mindfulness stress reduction program improves the quality of life of women in the menopausal period.
  Interventions: Other: mindfulness stress reduction program

INTERVENTIONS:
Other: mindfulness stress reduction program — mindfulness stress reduction program

SUMMARY:
The study was conducted to determine the effect of the mindfulness stress reduction program (MBSR) applied to postmenopausal women on menopausal complaints and quality of life. The population of the study was 2626 women and the sample was composed of 55 experimental and 63 control groups, totally 118 women. The data of the study were collected using Personal Information Form, Mindful Attention Awareness Scale (MAAS), Menopausal Symptoms Assessment Scale (MSAS) and Menopause Specific Quality of Life Scale (MYQOL).

DETAILED DESCRIPTION:
Aim: The study was conducted to determine the effect of the mindfulness stress reduction program (MBSR) applied to postmenopausal women on menopausal complaints and quality of life.

Materials and Methods: Research is quasi-experimental. The population of the study was 2626 women and the sample was composed of 55 experimental and 63 control groups, totally 118 women. The data of the study were collected using Personal Information Form, Mindful Attention Awareness Scale (MAAS), Menopausal Symptoms Assessment Scale (MSAS) and Menopause Specific Quality of Life Scale (MYQOL). In the study, an 8-week Mindfulness Stress Reduction Program was applied to the women in the experimental group. In the study, mid-test and post-test (MAAS, MSAS, MYQOL) were applied 8 and 16 weeks after the pre-test. Descriptive statistics, independent groups t test, chi-square test, ANOVA, Mauchly's test and Cronbach Alpha analysis were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

Being in menopause

* Not having any diagnosed psychiatric disease or using medication,
* Not using or not using hormone replacement therapy.

Exclusion Criteria:

* Having entered menopause with surgical methods,
* Not attending at least two group programs.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
mindfulness stress reduction program reduces menopausal symptoms | UP TO 16 WEEKS
  Menopause Rating Scale is an 11 item scale.The five-point Likert type scale has three sub-dimensions.The higher the scores of each item, the higher the complaints, the higher the total score of the scale, the higher the menopausal complaints.
Mindfulness stress reduction program improves quality of life | UP TO 16 WEEKS
  Menopausal Quality of Life Scale is a Likert-type scale with 29 questions and consists of four domains: vasomotor, psychosocial, physical and sexual. Each question score is from 0 to 6. The increase in the scale score indicates that the severity of the complaints increased.

CONTACTS AND LOCATIONS:
Locations (1):
- NURDİLAN, Elâzığ, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No